CLINICAL TRIAL: NCT06083324
Title: EXERT-C: Prospective Study of an EXErcise Regimen Designed to Improve Functional Mobility, Body Composition, and Strength After Treatment for Cancer
Brief Title: EXErcise Regimen Designed to Improve Functional Mobility, Body Composition, and Strength After Treatment for Cancer
Acronym: EXERT-C
Status: Recruiting | Type: Observational
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Colin Champ, MD, Radiation Oncologist, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Other Study IDs: 2023-021-SG
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: exercise; resistance training
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- General cancer patients: All patients undergoing treatment for cancer on an exercise regimen
  Interventions: Other: Dose escalated resistance training
- Head and neck cancer patients: All patients undergoing treatment for head and neck cancer on an exercise regime
  Interventions: Other: Dose escalated resistance training
- Colorectal cancer patients: All patients undergoing treatment for colorectal cancer on an exercise regime
  Interventions: Other: Dose escalated resistance training
- Pancreatic cancer patients: All patients undergoing treatment for pancreatic cancer on an exercise regime
  Interventions: Other: Dose escalated resistance training
- Metastatic breast cancer patients: All patients undergoing treatment for metastatic breast cancer on an exercise regime
  Interventions: Other: Dose escalated resistance training

INTERVENTIONS:
Other: Dose escalated resistance training — All individuals will be engaging in resistance training during and/or after their cancer treatment

SUMMARY:
This protocol seeks to analyze patient outcomes of the standard of care, monitored group exercise regimen of high-load resistance training and functional exercises with compound movements under close supervision on individuals who have been treated for cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-89 years
2. Women of child-bearing potential must verbally confirm lack of pregnancy prior to enrollment. They should also consent to use adequate contraception during the course of the study.
3. Participants must be determined capable of engaging in resistance training by exercise personnel and/or study PI
4. Participants must complete an assessment by EOC staff and be determined safe to engage in the workout regimen by the study exercise personnel.
5. Individuals not deemed safe to participate in the standard EOC exercise program will be referred to physical therapy or elsewhere

Exclusion Criteria:

1. Severe arthritic, joint, cardiovascular, or musculoskeletal condition that would interfere with exercise program

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with cancer on an exercise program at the AHN Exercise Oncology and Resiliency Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-01-26 (Estimated)

PRIMARY OUTCOMES:
Determine changes in fat mass in pounds from before to after the nutrition and exercise regimen via bioimpedance analysis | 3 months
  Measurement on bioimpedance analysis machine (Inbody 970)
Determine changes in fat mass in pounds from before to after the nutrition and exercise regimen via ultrasound | 3 months
  Measurement via ultrasound and calculation with Jackson-Pollack calculations
Determine changes in muscle mass in pounds from before to after the nutrition and exercise regimen | 3 months
  Measurement on bioimpedance analysis machine (Inbody 970)

SECONDARY OUTCOMES:
Determine changes in overall score of functional movement screen (FMS) from before to after the nutrition and exercise regimen | 3 months
  Determine changes in overall score of functional movement screen (FMS) from before to after the nutrition and exercise regimen
Determine changes in Y-balance score for each leg | 3 months
  Y-balance score adds up the distance each leg can move in the front and side directions, divided by the length of the hip. This correlates inversely with fall risk.
Determine changes in strength via load measured in pounds from before to after the nutrition and exercise regimen | 3 months
  Load is calculated by multiplying sets by repetitions by weight lifted for a specific exercise
Determine changes in EQ-5D responses 1-5 and overall score from before to after the nutrition and exercise regimen | 3 months
  EQ-5D asks 5 questions rates from 1-5 and an overall rating of health

CONTACTS AND LOCATIONS:
Locations (1):
- AHN CI Exercise Oncology and Resiliency Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Champ CE, Carpenter DJ, Diaz AK, Rosenberg J, Ackerson BG, Hyde PN. Resistance Training for Patients with Cancer: A Conceptual Framework for Maximizing Strength, Power, Functional Mobility, and Body Composition to Optimize Health and Outcomes. Sports Med. 2023 Jan;53(1):75-89. doi: 10.1007/s40279-022-01759-z. Epub 2022 Sep 29. PMID 36175646